CLINICAL TRIAL: NCT01561456
Title: Phase II, Randomized, Open-label Study of the IGF-1R Inhibitor AXL1717 Compared to Docetaxel in Patients With Previously Treated, Locally Advanced, or Metastatic Squamous Cell Carcinoma or Adenocarcinoma of the Lung
Brief Title: Study of AXL1717 Compared to Docetaxel to Treat Squamous Cell Carcinoma or Adenocarcinoma of the Lung
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Axelar AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AXL-003; 2011-002007-15 (EudraCT Number)
Record Dates: First submitted 2012-03-05; First posted 2012-03-23 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-12

CONDITIONS: Non-small-cell Lung Cancer; Squamous Cell Carcinoma; Adenocarcinoma of the Lung
Keywords: non-small-cell lung cancer; squamous cell carcinoma; adenocarcinoma of the lung; IGF-1 inhibitor; docetaxel; AXL1717; NSCLC; SCC; AC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Squamous Cell; Adenocarcinoma of Lung | interventions — picropodophyllin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AXL1717 (Experimental): AXL1717
  Interventions: Drug: AXL1717
- Docetaxel (Active Comparator): Docetaxel
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: AXL1717 — AXL1717 administered as oral suspension at 400 mg twice daily for 21 days per cycle; i.e. daily for up to four cycles
  Other Names: small molecule IGF-1 inhibitor
  Arms: AXL1717
Drug: Docetaxel — Docetaxel administered as a standard treatment (75 mg/m2 IV infusion over 1 hour) once every three weeks throughout the 4-cycle study
  Other Names: Taxotere
  Arms: Docetaxel

SUMMARY:
The purpose of this study is to compare effectiveness and safety of experimental anticancer medicine, AXL1717, and docetaxel in patients with squamous cell carcinoma or adenocarcinoma of the lung.

DETAILED DESCRIPTION:
Non-Small-Cell lung Cancer (NSCLC) is the most common form of lung cancer, and treatment with cytotoxic chemotherapy only provides a 10% reduction in the risk of death in patients with advanced NSCLC. One-third of all non-resectable advanced NSCLC patients in second line do not receive chemotherapy treatment at all. In the absence of treatment the Progression-Free Survival (PFS) for NSCLC patients is dismal, in the range of 6-8 weeks, and treatment only modestly improves the median PFS to 10-11 weeks. Therefore, because of an overall poorer prognosis for patients with advanced NSCLC, development of new agents is urgently needed.

AXL1717 is a small molecule experimental product developed by Axelar AB as anticancer agent for oral administration. AXL1717 inhibits the insulin-like growth factor 1 (IGF-1), which is often over expressed in lung tumors and can mediate the proliferation of lung cancer cells and resistance to therapy. Results of previous preclinical and clinical studies indicate that AXL1717 will be tolerable and effective in patients with previously-treated, advanced squamous cell carcinoma (SCC) and adenocarcinoma (AC) histological subtypes of NSCLC.

This is an open label, randomized, multi-center, Phase II study to investigate AXL1717 compared to docetaxel in patients with squamous cell carcinoma (SCC) or adenocarcinoma (AC) of the lung. Patients with previously treated, locally advanced or metastatic SCC or AC subtypes of NSCLC in need of additional treatment will be enrolled in the study. Patients will be randomized to either AXL1717 or to docetaxel group as monotherapy, in a 3:2 ratio for each NSCLC subtype. Patients in AXL1717 group will receive 400 mg AXL1717 twice daily (BID) as oral suspension for 21 days per cycle; i.e. daily for up to four cycles unless a dose interruption, delay, or reduction is required. Docetaxel will be administered as a standard treatment (75 mg/m2 IV infusion over 1 hour) once every three weeks throughout the 4-cycle study. The primary objective of the study is to compare the rate of progression-free survival (PFS) at 12 weeks between patients treated with AXL1717 and patients treated with docetaxel. Additional efficacy and safety parameters will be monitored throughout the study. Patients treated with AXL1717 who are responding to treatment or remain stable at the end of 4 cycles may be offered an extension of treatment with AXL1717.

ELIGIBILITY:
Inclusion Criteria:

* informed of the study and have provided written informed consent
* At least 18 years of age
* Histologically confirmed diagnosis of locally advanced, or metastatic squamous cell carcinoma or adenocarcinoma histological subtypes of non-small-cell lung cancer (stage IIIB or IV)
* For patients with squamous cell histology: previously treated with first-line chemotherapy and has had disease progression during or after first-line therapy.
* For patients with adenocarcinoma histology: previously treated with one or two lines of chemotherapy.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy ≥ 3 months
* Measurable disease by RECIST 1.1 criteria
* Hematology values: blood leukocyte count ≥ 3.0 x 109/L, blood absolute neutrophil count ≥ 1.5 x 109/L, blood platelet count ≥ 100 x109/L, hemoglobin ≥ 100 g/L (transfusions are allowed)
* Clinical chemistry values: plasma total bilirubin level ≤ upper limit of the "normal" range (ULN; i.e. reference), plasma AST or ALT ≤ 1.5 x ULN (≤ 5 times if liver metastases have been documented) and plasma creatinine ≤ 2.0 x ULN
* 12-lead ECG with normal tracings

Exclusion Criteria:

* Mixed histology of squamous and non-squamous NSCLC
* Ongoing infection or other major recent or ongoing disease that, according to the Investigator, poses an unacceptable risk to the patient
* Known primary or secondary central nervous system malignancy.
* Active or previously treated carcinomatous meningitis
* Truly non-measurable disease by RECIST 1.1 criteria, such as patients with one or more of the following without any RECIST measurable disease:

  * Bone lesions
  * Ascites
  * Pleural or pericardial effusion
  * Lymphangitis cutis or pulmonis
  * Cystic lesions
* Grade 3 or higher constipation within the past 28 days or grade 2 constipation within the past 14 days before randomization.
* Active hepatitis B, active hepatitis C, or known HIV infection
* Coexisting uncontrolled medical condition, including active cardiac disease (such as unstable angina, myocardial infarction within 6 months, or New York Heart Association Class III/IV congestive heart failure), and significant dementia
* Hepatic impairment as indicated by abnormalities of transaminases (AST and/or ALT > 1.5 × ULN or AST and/or ALT > 5 times ULN if liver metastases have been documented) and/or increased alkaline phosphatase (> 2.5 × ULN) considered as a result of hepatic impairment (and not from bone disease)
* History of cancer that has required treatment or been active within the past 5 years, other than NSCLC, basal cell carcinoma, or cervical carcinoma in situ
* Major surgical procedure within 4 weeks prior to randomization
* More than one prior anti-tumor systemic therapy for advanced squamous cell NSCLC, and more than two prior lines of chemotherapy for advanced adenocarcinoma NSCLC
* Previous use of docetaxel in any line of therapy
* Women of child bearing potential (WOCBP) who do not consent to using acceptable methods of contraception
* Women who are breast-feeding or have a positive pregnancy test at screening
* Current participation in any other investigational clinical trial or any administration of an investigational agent within 4 weeks of study drug administration
* ECOG performance status > 2
* Life expectancy < 3 months
* Known or suspected hypersensitivity to AXL1717 or docetaxel or to drugs formulated with polysorbate 80
* Lack of suitability for participation in the trial, for any reason, as judged by the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Rate of progression-free survival (PFS) | 12 weeks

SECONDARY OUTCOMES:
Rate of complete response (CR), partial response (PR), stable disease, (SD), progressive disease (PD), disease control (CR + PR + SD), and objective response (CR + PR) | 12 weeks
Median time to disease progression (TTP), time to objective response and time to treatment failure (TTF) | 17 weeks
Median duration of progression-free-survival (PFS), objective response and disease control | 17 weeks
12-week survival | 12 weeks
1 year survival | 1 year
Investigational product toxicity profile | 17 weeks
Overall survival | time from randomization to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bergqvist, MD, PhD, Principal Investigator — Uppsala University Hospital, Sweden
Locations (24):
- Belarus (4):
  - State Medical Institution: Republic Scientific Oncology Center, Poselok, Minsk Oblast
  - Gomel Regional Clinical Oncology Center, Homyel
  - Minsk City Clinical Oncology Center, Minsk
  - Vitebsk Regional Clinical Oncology Center, Vitebsk
- Hungary (4):
  - Semmelweis University; Clinic for Pulmonology, Budapest
  - University of Debrecen Medical and Health Science Center, Clinic of Pulmonology, Debrecen
  - Kenezy Gyula County Hospital, Debrecen
  - Hospital for Thoracic Diseases of Csongrad County Local Government, Deszk
- Poland (2):
  - Wladyslaw Bieganski Regional Specialist Hospital, Grudziądz
  - Maria Sklodowska-Curie Institute of Oncology in Warsaw, Warsaw
- Russia (7):
  - State Therapeutical and Prophylactic Institution: Chelyabinsk Regional Oncology Center, Chelyabinsk
  - City Clinical Hospital #1, Novosibirsk
  - Orel Oncology Center, Oryol
  - St. Petersburg State Medical Institution Municipal Clinical Oncology Center, Saint Petersburg
  - State Higher Educational Institution St. Petersburg State Medical University n. a. after I. P. Pavlov under Federal Agency for Healthcare and Social Development, Research Institute of Pulmonology, Saint Petersburg
  - Tula Regional Oncology Center, Tula
  - Sverdlovsk Regional Oncology Center, Yekaterinburg
- Ukraine (7):
  - Dnipropetrovsk City Multispecialty Clinical Hospital #4, Dniepropetrovsk
  - Public Clinical Treatment and Prophylaxis Institution: Donetsk Regional Antitumor Center, Donetsk
  - Kharkiv, State Institution: S.P. Hryhoriev Institute of Medical Radiology under the Ukrainian Academy of Medical Sciences, Kharkiv
  - Public Healthcare Institution: Kharkiv Regional Clinical Oncology Center, Kharkiv
  - Kyiv City Oncology Hospital, Kyiv
  - Lviv State Regional Treatment and Diagnostics Oncology Center, Lviv
  - Zakarpattia Regional Clinical Oncology Center, Uzhhorod